CLINICAL TRIAL: NCT00252278
Title: The Effect of a Once Daily Evening Dose of Atomoxetine (ATX) on ADHD-Related Insomnia in Children and Adolescents
Brief Title: Effect of Atomoxetine on ADHD-Related Insomnia in Children and Adolescents
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0120-05
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2006-07-07 (Estimated); Status verified 2005-11

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD); Insomnia
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Sleep Initiation and Maintenance Disorders | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: atomoxetine

SUMMARY:
Children and adolescents with Attention-Deficit/Hyperactivity Disorder (ADHD) very commonly experience difficulty in initiating and maintaining sleep. Studies have shown that daytime sleepiness resulting from insufficient sleep can affect attention and learning. Therefore, treating insomnia in children with ADHD may not only improve sleep, but it could potentially improve ADHD symptoms as well.

The main purpose of this study is to examine the effects of atomoxetine on ADHD-related insomnia. Atomoxetine (Strattera®) is a non-stimulant drug used to treat ADHD symptoms in both children and adults, and there is evidence that it may also have a positive effect on sleep in children with ADHD. During the study, participants will receive either atomoxetine or placebo for a period of four weeks. We expect that the effects of atomoxetine on sleep will differ from those of placebo, with atomoxetine having a greater effect on improving sleep difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Boy or girl aged 6-17 years, inclusive, and English-speaking
* Meet the DSM-IV criteria for Attention-Deficit/Hyperactivity Disorder
* Have sleep initiation defined by:

  1. difficulty initiating or maintaining sleep that is viewed as a problem by the child or caregiver
  2. sleep onset delay that is not exclusively related to direct or rebound effects of psychostimulant treatment
* Have a parent or legal guardian willing to participate in the study

Exclusion Criteria:

* Have any other primary sleep disorder(s) (e.g. obstructive sleep apnea or periodic limb movement disorder)
* Have a history of significant chronic medical (e.g. diabetes, severe asthma) or psychiatric (e.g. depression) illness
* Have a history of chronic use of sedating (e.g. antihistamines) or alertness enhancing (e.g. caffeine) medications
* Have a history of failure to respond to an adequate (defined as appropriate dose and adequate duration of therapy) previous trial with atomoxetine

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36
Dates: Start 2005-11

PRIMARY OUTCOMES:
mean sleep onset latency
parent and child-reported evening settling difficulties

SECONDARY OUTCOMES:
night wakings, sleep duration, and sleep efficiency
daytime sleepiness
ADHD symptom improvement
executive functions and functional outcomes/quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Judith Owens, MD, MPH, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States